CLINICAL TRIAL: NCT01064869
Title: Evaluation of the Benefits of an Individualised Menu Driven Nurse Led Programme to Improve Adherence in Difficult Asthma
Brief Title: A Nurse Led Programme to Improve Adherence in Difficult Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Liam Heaney, Doctor, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 05/NIR/03/32
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Adherence; Asthma; medication
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycho-educational intervention (Experimental): A nurse-led programme of intervention will be devised. Patients will attend weekly for a period of 12 weeks. It will have two stages incorporating:
  1. Structured interview to identify demographic information and individual reasons for non-adherence and assessment of readiness to change behaviour
  This will be followed by an individualised package incorporating:
  1. A structured asthma education programme, to address any gaps in asthma knowledge or requests for information
  2. Motivational interviewing based on stages of change model to encourage change and adherence
  3. Psychological therapy involving (a) relaxation therapy (b) cognitive behavioural techniques looking at negative and catastrophic thoughts and (c) panic cycle adapted to respiratory patients
  Interventions: Behavioral: Pyscho-behavioural
- usual care (No Intervention): Standard asthma management

INTERVENTIONS:
Behavioral: Pyscho-behavioural — A nurse-led programme of intervention will be devised. Patients will attend weekly for a period of 12 weeks. It will have two stages incorporating:
  1. Structured interview to identify demographic information and individual reasons for non-adherence and assessment of readiness to change behaviour
  This will be followed by an individualised package incorporating:
  1. A structured asthma education programme, to address any gaps in asthma knowledge or requests for information
  2. Motivational interviewing based on stages of change model to encourage change and adherence
  3. Psychological therapy involving (a) relaxation therapy (b) cognitive behavioural techniques looking at negative and catastrophic thoughts and (c) panic cycle adapted to respiratory patients
  Arms: Psycho-educational intervention

SUMMARY:
Approximately 5% of adults with asthma have difficult to control disease but these account for up to 80% of total cost of asthma due to recurrent healthcare contact including hospital admission. The reasons for "difficult asthma" are multi-factorial, but an important element in many patients is non-adherence to steroid therapy. Recent qualitative analysis by the investigators group has identified a number of both individual and group themes, related to non-adherence with steroid treatment. Many of these themes such as steroid phobia, inaccurate / lack of knowledge, negative attitudes and inability to deal with side-effects, are potentially modifiable and the investigators believe, unless these issues are addressed, at an individual patient level, adherence is unlikely to improve. This randomised parallel group study will examine a nursing intervention to try and improve adherence and as a consequence, asthma control, in a group of difficult asthmatics where non-adherence has been identified as a significant factor. The study will use a needs-led menu driven individualised intervention and will compare this to current best asthma care. The primary outcome measure will be adherence to therapy, however asthma control, lung function and asthma related quality of life, patients' attitudes to asthma and treatment and their levels of anxiety and depression will also be examined. Addressing the issue of non-adherence is fundamental to improving asthma management in this difficult group with concomitant reduction on health care costs and improvements in patients' quality of life

DETAILED DESCRIPTION:
Plan of investigation The study will be a single blind randomised controlled trial. Patients will be recruited from those attending the difficult asthma clinic at the Belfast City Hospital and deemed non-adherent (see below). Difficult asthma will be defined as; 1. persisting asthma symptoms (Asthma control score >3)(ACS), despite detailed assessment and management; 2. minimal maintenance therapy of long acting B2-agonist and inhaled steroids ( 800 mcg BDP or equivalent) and 3. at least 1 course of systemic steroids in the preceding 12 months.

Non adherence will be defined as prescription filling of <50% of prescribed anti-inflammatory inhaled therapy utilized in preceding 6 months (from GP prescription records). All subjects will be invited to take part and give consent to take part in the study.

Exclusion criteria will be medication adherence, a condition other than asthma contributing to persisting symptoms; current smoker; significant co-morbidity due to condition other than asthma. Primary Outcome measure Improvement in adherence to steroid therapy before and after intervention (both 7 day prednisolone (serum assay) and inhaled steroid therapy (prescription counting).

Secondary outcome measures Improvement in Asthma Control Scores (ACS) Improvement in asthma Quality of Life Questionnaire (AQLQ) Improvement in Lung function Reduction in courses of rescue steroid Hospital Anxiety and Depression Scale These are all routinely measured as part of the difficult asthma service. Study design Pre run-in period

1. Assessment of inclusion / exclusion criteria
2. Full informed consent Run-in period (1 week)- All participants Week 1 Prednisolone course - 7 day course

1. ACS/Forced expiratory volume in 1 second (FEV1) on Day 1 (Lung function breathing test) 2. Serum prednisolone/cortisol and urinary cortisol/creatinine ratio on Day 7 - measures adherence to prednisolone 3. Asthma control score/FEV1 Day 7 Randomisation Patients will be randomized into two groups either control (usual care) or intervention group using a random number generator.

Intervention

Intervention Group- A nurse-led programme of intervention will be devised. It will have two stages incorporating:

1. Semi-structured audio taped interview to identify individual reasons for non-adherence and assessment of readiness to change behaviour.
2. An individualised package incorporating:

   1. Asthma education programme to address any specific gaps in asthma knowledge or requests for information
   2. Motivational interviewing based on stages of change model to encourage change and adherence
   3. Psychological therapy involving (a) relaxation therapy (b) cognitive behavioural techniques looking at negative and catastrophic thoughts and (c) panic cycle adapted to respiratory patients Patients will be seen regularly (individual needs determine time spans) for a period of 3 months.

Control group - standard asthma management. Outcome measures Primary outcome measures Adherence will be determined at baseline, 3 and 9 months by prescription filling to define outcome after completion of programme. During the period of follow-up, when a further 7 day course of prednisolone is indicated on clinical grounds, serum prednisolone/cortisol and urinary cortisol/creatinine ratio will be measured on completion of course.

Secondary outcome measures These will be measured at 3 and 9 months There are currently 200 patients attending the difficult asthma service at Belfast City Hospital Trust all of whom fulfil our definition of difficult asthma. No data is available in this specific population regarding adherence with inhaled therapy but based on adherence with prednisolone and adherence data with inhaled therapy in other severities of asthma, we would anticipate that over 50% will be variably adherent to therapy. 1-6 months - Screening population / liaising with primary care / psychological intervention training 6 months-18 months - Patient recruitment and intervention package delivered 18-36 months- Follow-up and data analysis.

ELIGIBILITY:
Inclusion Criteria:

Filling <50% of prescription refills for inhaled combination therapy

* Persisting asthma symptoms (ACS >3) despite detailed assessment and management
* Minimal maintenance therapy of long acting beta2-agonist and inhaled steroids (800mg BDP or equivalent)
* At least 1 course of systemic steroids in the preceding 12 months.

Exclusion Criteria:

Medication adherence

* A condition other than asthma contributing to persisting symptoms
* Current smoker
* Ex-smoker > 10 pack years -Significant co-morbidity due to condition other than asthma.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Adherence to Inhaled combination therapy | 6 months

SECONDARY OUTCOMES:
Asthma control score | 6 months
Asthma Quality of Life Questionnaire | 6 months
Hospital anxiety and depression scale | 6 months
Lung function | 6 months
Reduction in rescue courses of Steroids | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Liam Heaney, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Regional Respiratory Centre, Belfast City Hospital, Belfast, Co Down, United Kingdom